CLINICAL TRIAL: NCT05928052
Title: Transcutaneous Spinal Cord Stimulation to Improve Respiratory Function and Shorten Ventilator Dependence in Patients with ARDS
Brief Title: Spinal Cord Stimulation to Shorten Ventilator Dependence in ARDS Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Daniel Lu, MD, PhD, Professor, Neurosurgery, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 21-001220
Record Dates: First submitted 2023-05-23; First posted 2023-07-03 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Respiratory Distress Syndrome
Keywords: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ARDS cohort (Experimental): Patient diagnosed with ARDS. Treated daily for 60 minutes with transcutaneous cervical and/or thoracic spinal stimulation
  Interventions: Device: Transcutaneous Biopac Electrical Stimulator
- Surgery Cohort (Active) (Experimental): Patient undergoing inpatient non-cardiac surgery admitted to the intensive care unit (ICU) after surgery. Treated daily for 60 minutes with transcutaneous cervical and/or thoracic spinal stimulation
  Interventions: Device: Transcutaneous Biopac Electrical Stimulator

INTERVENTIONS:
Device: Transcutaneous Biopac Electrical Stimulator — A transcutaneous electrical stimulator sends low levels of electrical current through surface hydrogel electrodes directly to the spinal cord to improve function.

SUMMARY:
This is an early phase, proof-of-concept clinical trial assessing the safety and feasibility of non-invasive spinal cord stimulation to prevent respiratory muscle atrophy in mechanically ventilated ARDS patients. The investigators will recruit 10 elective surgery patients (surgery cohort) and 10 ARDS patients (ARDS cohort) for this study. A non-invasive, alpha-prototype Restore Technology stimulator using hydrogel surface electrodes will be used to stimulate the spinal cord at the cervical or thoracic level.

DETAILED DESCRIPTION:
Stimulation will be conducted in closed-loop fashion at the start of inspiratory cycle. Signal from a chest belt will be used to synchronize stimulation with ventilator and prevent interference with ventilator (see Protection of Human Subjects). Prior to treatment stimulation, mapping will be conducted at 1 Hz with electrodes placed in locations identified to be optimal in the surgery cohort. Assessment of evoked EMG responses from respiratory muscles will be conducted. Once this electrode configuration is confirmed as effective (capable of evoking EMG activity), stimulation with this configuration will be applied for treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18-85 years;
2. Intubated with confirmed diagnosis of ARDS (by Berlin Criteria: acute onset within one week of known insult, bilateral airspace opacities not fully explained by pleural effusions, atelectasis, and/or nodules, respiratory failure not explained by heart failure or fluid overload, PaO2/FiO2 ratio < 300); or identified as a patient admitted to the intensive care unit (ICU) after non-cardiac surgery;
3. Able to provide informed consent or available next of kin able to provide informed consent;
4. Have intact chest/lung, upper and lower extremity anatomy;
5. The neuromuscular connections between the spinal cord, diaphragm, and intercostal muscles are intact;
6. Enrollment of subject within 48 hours of intubation;
7. Able to induce evoked response of diaphragm muscle by spinal cord TES.

Exclusion Criteria:

1. Phrenic nerve or diaphragm pacer;
2. History of seizure disorder or on anti-epileptic medication for the treatment of seizures;
3. Compromised skin in back (neck, upper and lower back);
4. Pregnancy;
5. Implanted devices: cardiac pacemakers, implanted defibrillators, implanted neurostimulators, phrenic nerve pacers;
6. BMI greater than or equal to 35;
7. Pharmacological paralysis/neuromuscular blockade*.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2027-01-06 (Estimated); Study Completion 2029-01-06 (Estimated)

PRIMARY OUTCOMES:
Recording of significant stimulation-induced adverse events (AE) | 1-48 months
  Although unlikely, we will record and monitor the number of stimulation-induced adverse events per case and per cohort. Our goal is to have an overall AE rate of less than 10% per cohort.

SECONDARY OUTCOMES:
Recording of total ventilation time | 1-48 months
  The total time that patient is ventilated will be recorded to determine if stimulation reduces total intubation time
Measurement of diaphragm thickness | 1-48 months
  Evidence of maintenance of diaphragm muscle thickness (in mm) by ultrasound
Assessment of diaphragm and respiratory muscle EMG amplitudes | 1-48 months
  EMG amplitudes of diaphragm and other muscles involved in respiration (intercostals, trapezius, abdominal) will be measured at a couple time points throughout the study period to determine if stimulation can maintain muscle response.
Measurement of respiratory pressure | 1-48 months
  Peak Inspiratory and Expiratory pressure measurements (in mm Hg) will be recorded from ventilation units to determine if stimulation maintains or improves respiratory airway pressure.
Assessment of respiratory tidal volume | 1-48 months
  Respiratory Tidal Volume (voluntary and resting) will be recorded (in mL) to determine if stimulation assists in maintaining or improving lung capacity.
Measurement of ventilator weaning time | 1-48 months
  Measurements of ventilator weaning time will be recorded to determine if stimulation assists in decreasing the total time from complete intubation to complete extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lu, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UCLA Clinical Trials — https://www.uclahealth.org/clinical-trials